CLINICAL TRIAL: NCT01888081
Title: Phase I/II Trial of A-dmDT390-bisFv(UCHT1) Fusion Protein in Combination With Ionizing Radiation for the Treatment of Stage IV Melanoma
Brief Title: A-dmDT390-bisFv(UCHT1) Fusion Protein in Combination With Ionizing Radiation for Treatment of Stage IV Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Protocol replaced with combination therapy adding KEYTRUDA (pembrolizumab)
Sponsor: Angimmune LLC (Industry)
Collaborators: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCC-MEL-13
Record Dates: First submitted 2013-06-21; First posted 2013-06-27 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Radiation, Ionizing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A-dmDT390-bisFv(UCHT1) with Ionizing Radiation (Experimental): A-dmDT390-bisFv(UCHT1) Fusion Protein in Combination With Ionizing Radiation
  Interventions: Drug: A-dmDT390-bisFv(UCHT1) (Resimmune®); Radiation: Ionizing Radiation

INTERVENTIONS:
Drug: A-dmDT390-bisFv(UCHT1) (Resimmune®)
Radiation: Ionizing Radiation

SUMMARY:
The purpose of this trial is to study A-dmDT390-bisFv(UCHT1) in combination with ionizing irradiation for the treatment of stage IV melanoma, a disease that is essentially incurable with median overall survival periods that range from 8-16 months.

DETAILED DESCRIPTION:
A-dmDT390-bisFv(UCHT1) (Resimmune™), an anti-T cell immunotoxin is currently being studied as a treatment for cutaneous T cell lymphoma and other CD3+ malignant diseases (FDA IND Number: 100712, Scott and White Protocol 071163). During the course of this study, data accumulated that Resimmune could be acting as an immunomodulator. This was based on the observation that four out of six partial responses converted to complete responses at times ranging between 6 and 24 months following the completion of the 4-day treatment protocol and no other treatment took place.

The purpose of this trial is to test the hypothesis that Resimmune can act as an immunomodulator of late stage metastatic melanoma when combined with palliative radiation to induce the priming of activated T cells with tumor antigens. The primary objective of this study is to determine the safety of combining Resimmune with palliative radiation therapy in patients with stage IV melanoma. A secondary objective is to document the tumor response and duration of response at irradiated and unirradiated sites (the abscopal effect). An additional secondary objective is to determine if T cell activation occurs following administration of A-dmDT390-bisFv(UCHT1) and local radiation to a metastatic lesion of melanoma.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically proven stage IV metastatic melanoma consisting of at least two lesions
* Patients must have a performance status of < 2 on Eastern Cooperative Oncology Group scale (see Appendix).
* Patients must have bilirubin < 1.5 mg/dL, transaminases < 2.5 X ULN, albumin > 3 gm/dL, creatinine < 2.0 mg/dL, adequate pulmonary function by physical exam and pulse oximetry and adequate cardiac reserve (EF > 50% normal). Patients must have a normal echocardiogram without any evidence of cardiac chamber hypertrophy, dilatation or hypokinesis.
* Patients must give written informed consent prior to registration.
* Females and males must be willing to use an approved form of birth control while on this study and for 2 weeks after completion.
* Patients of ages 18-80 are eligible provided they have stage IV melanoma and are negative for BRAF or have failed BRAF inhibitor treatment or if they have failed or are intolerant to other established therapy known to provide clinical benefit for their condition or if they have been adequately consented and agreed to forgo FDA approved clinically meaningful therapy

Exclusion Criteria:

* Inability to give informed consent because of psychiatric problems, or complicated medical problems.
* Serious concurrent medical problems, uncontrolled infections, or disseminated intravascular coagulopathy (DIC).
* Preexisting cardiovascular disease, the only exception being well controlled essential hypertension with a sitting blood pressure of <155 systolic and <90 diastolic without any evidence of structural heart disease or one episode of myocardial infarction > 8 months ago. A past history of the any of the following are exclusions: congestive heart failure, atrial fibrillation, pulmonary hypertension, anticoagulant drug therapy, thromboembolic events, cardiomyopathy or a myocardial infarction within the past 8 months.
* Pregnant or nursing women will be excluded from study.
* History of congestive heart failure.
* History of cirrhosis of the liver

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-02; Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Immune-related overall response rate (irORR) | For up to 1 year post treatment or until disease progression
  Response will be assessed at 2 months, and at least every 3 months (±7 days) thereafter using for up to 1 year after the last treatment administration or until evidence of disease progression. Tumor measurements and therapeutic response will be determined using irRC (Immune Related Response Criteria). At a minimum, CT scans of the chest, abdomen, and pelvis will be performed at study entry, at 2 months, and, if a response or stable disease, at least every 3 months (±7 days) for up to 1 year after the last dose of study drug, and/or at any time there is clinical evidence of disease progression, to evaluate disease status.

SECONDARY OUTCOMES:
Overall survival | every 3 months for up to 3 years
  Survival should be assessed and a physical exam should be completed every three months as per standard of care

OTHER OUTCOMES:
Treatment Duration | 4 Days
  Patients will be admitted to the hospital on day 0 for the first two infusions on day 1. Infusions for days 2, 3 and 4 and fractionated radiation will be done in the clinic on an outpatient basis.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chesney, MD, PhD, Principal Investigator — James Graham Brown Cancer Center, University of Louisville
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States